CLINICAL TRIAL: NCT00582140
Title: Phase I Study of a DNA-based Vaccine Targeting Prostatic Acid Phosphatase (PAP) in Patients With Stage D0 Prostate Cancer
Brief Title: Prostatic Acid Phosphatase (PAP) Vaccine in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0365; CO04806 (Other: University of Wisconsin Carbone Cancer Center); DOD-A-13390 (Other: DOD); A534260 (Other: UW Madison); SMPH/MEDICINE (Other: UW Madison); 2004-0365 (Other: Institutional Review Board)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2015-07

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Stage D0; Non-Metastatic; Rising PSA
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — regramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort Level 1 (Experimental): pTVG-HP (dose 1: 100 μg) with rhGM-CSF (200 μg); administered i.d. biweekly for 6 total doses
  Interventions: Biological: pTVG-HP with rhGM-CSF
- Cohort Level 2 (Experimental): pTVG-HP (dose 2: 500 μg) with rhGM-CSF (200 μg); administered i.d. biweekly for 6 total doses
  Interventions: Biological: pTVG-HP with rhGM-CSF
- Cohort Level 3 (Experimental): pTVG-HP (dose 3: 1,500 μg) with rhGM-CSF (200 μg); administered i.d. biweekly for 6 total doses
  Interventions: Biological: pTVG-HP with rhGM-CSF

INTERVENTIONS:
Biological: pTVG-HP with rhGM-CSF — pTVG-HP (dose 1: 100 μg) with rhGM-CSF (200 μg); administered i.d. biweekly for 6 total doses
  Arms: Cohort Level 1
Biological: pTVG-HP with rhGM-CSF — pTVG-HP (dose 2: 500 μg) with rhGM-CSF (200 μg); administered i.d. biweekly for 6 total doses
  Arms: Cohort Level 2
Biological: pTVG-HP with rhGM-CSF — pTVG-HP (dose 3: 1,500 μg) with rhGM-CSF (200 μg); administered i.d. biweekly for 6 total doses
  Arms: Cohort Level 3

SUMMARY:
The investigators are trying to find new methods to treat prostate cancer. The approach they investigators are taking is to try to enhance patients own immune response against the cancer. In this study the investigators will be testing the safety of a vaccine that may be able to help the body fight prostate cancer.

DETAILED DESCRIPTION:
The purpose of this research is to determine the safety of serial intradermal vaccinations of a DNA vaccine encoding human PAP, with GM-CSF as a vaccine adjuvant, in subjects with stage D0 prostate cancer. In addition, to determine whether PAP-specific IFNУ-secreting CD8+ T cells can be augmented in subjects with stage D0 prostate cancer by means of immunization with a plasmid DNA vaccine encoding PAP.

This is a phase I design where patients will receive the vaccine pTVG-HP with rhGM-CSF administered i.d. biweekly for 6 total doses. There will be three escalating dose cohorts. The dosing cohort considered to be the maximum tolerated dose level will be expanded up to a total of 16 patients.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologic diagnosis of adenocarcinoma of the prostate
* Must have completed local therapy by surgery and/or ablative radiation therapy at least 2 months prior to entry.
* Must have clinical stage D0 disease defined by the following: In patients treated by surgery, serum PSA values must be > 2 ng/ml by two measurements at least two weeks apart. In patients treated with ablative radiation therapy, three consecutive increases in serum PSA must be documented, with at least a one month interval between values with the finalPSA > 2ng/ml.
* Prior history of a second malignancy is allowed if treated with curative intent disease free for > 5 years.
* Karnofsky performance score of > 70

Exclusion Criteria:

* No evidence of immunosuppression or have been treated with immunosuppressive therapy, such as chemotherapy, chronic treatment dose corticosteroids (greater than the equivalent of 10 mg prednisone per day), or radiation therapy to >30% of the bone marrow, within 6 months of the first vaccination.
* Must not be on concurrent androgen ablative (hormonal) therapy, or must have completed this therapy at least one month prior to study entry.
* Must not have demonstrated PSA progression during any prior hormonal therapy or chemotherapy.
* Must not have known evidence of bone metastases or non-regional lymph node involvement (stage D2 disease) as determined by bone scan or CT scan. -Must not have been treated previously with another investigational anti- tumor vaccine.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this phase I study is to determine if the vaccination with serial intradermal vaccinations of a DNA-based vaccine targeting PAP, with GM-CSF is safe (the investigators will be evaluating the degree of toxicity seen) | During study treatment and for 15 year follow-up
To determine whether PAP-specific IFNγ-secreting CD8+ T cells can be generated in patients with stage D0 prostate cancer by means of immunization with a plasmid DNA vaccine encoding PAP. | 12 months

SECONDARY OUTCOMES:
Efficacy: Immune Response and PSA response | During treatment and one year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Johnson LE, Olson BM, McNeel DG. Pretreatment antigen-specific immunity and regulation - association with subsequent immune response to anti-tumor DNA vaccination. J Immunother Cancer. 2017 Jul 18;5(1):56. doi: 10.1186/s40425-017-0260-3. PMID 28716080
- [Derived] Tonelli TP, Eickhoff JC, Johnson LE, Liu G, McNeel DG. Long-term follow up of patients treated with a DNA vaccine (pTVG-hp) for PSA-recurrent prostate cancer. Hum Vaccin Immunother. 2024 Dec 31;20(1):2395680. doi: 10.1080/21645515.2024.2395680. Epub 2024 Aug 29. PMID 39208856
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu